CLINICAL TRIAL: NCT07069465
Title: Pilot Study to Determine the Effect of Androgen Deprivation Therapy on the Sensitivity of PSMA-PET Scanning for Patients Undergoing Initial Staging Prior to Robot-Assisted Laparoscopic Radical Prostatectomy and Pelvic Lymphadenectomy
Brief Title: Pilot Study: Androgen Deprivation Therapy Impact on PSMA-PET Sensitivity in Prostatectomy Staging
Acronym: PIONEER PSMA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Urology Clinics of North Texas (Network)
Collaborators: Blue Earth Diagnostics (Industry); Texas Health Resources (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU-2023-1275
Record Dates: First submitted 2024-05-29; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate, Prostate Cancer, Androgen Deprivation Therapy, Posluma, Orgovyx, PSMA-PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Active Comparator): 5 patients (Cohort A) undergo a second study PSMA-PET with POSLUMA® 3 weeks after initiation of ADT and discontinue ADT immediately after the scan is completed.
  Interventions: Diagnostic Test: flotufolastat F 18; Drug: Relugolix 120 MG; Diagnostic Test: Serum PSA and Testosterone
- Cohort B (Active Comparator): 5 patients (Cohort B) undergo a second study PSMA-PET with POSLUMA® 6 weeks after initiation of ADT and discontinue ADT immediately after the scan is completed.
  Interventions: Diagnostic Test: flotufolastat F 18; Drug: Relugolix 120 MG; Diagnostic Test: Serum PSA and Testosterone

INTERVENTIONS:
Diagnostic Test: flotufolastat F 18 — PSMA-PET scan with Posluma agent (x2)
  Other Names: Posluma
Drug: Relugolix 120 MG — Administration of oral ADT for 3 and 6 weeks
  Other Names: Orgovyx
Diagnostic Test: Serum PSA and Testosterone — Serum PSA and testosterone at study initiation and again at 3 and 6 weeks after initiation of ADT

SUMMARY:
This is a pilot, non-randomized, two-cohort interventional study in patients who meet the inclusion criteria, using an FDA- approved androgen deprivation agent for a 3 or 6-week course of treatment prior to standard-of-care RALP with PLND. The intent of the study is to determine the effect of ADT on PSMA expression as measured by PSMA-PET scan. A second PSMA-PET scan will be performed after ADT for either 3 or 6 weeks, depending on cohort, prior to RALP and PLND.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with unfavorable intermediate or high-risk prostate cancer where RALP and PLND is planned and consulted with primary urologist

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
1. Mean change in maximum standardized uptake value (SUVmax) per lesion as measured by PSMA-PET (POSLUMA®) from baseline to post-ADT | 3-6 weeks
  Time Frame: Baseline and 3-6 weeks after initiation of ADT Description: SUVmax will be measured on PSMA-PET for each lesion identified prior to ADT and again after 3 or 6 weeks of ADT (depending on cohort). The primary metric will be the mean change in SUVmax per lesion, per participant. Data will be summarized as mean ± SD, and analyzed using paired statistical testing to determine significance of change.
New lesions not identified pre-treatment are detectable after ADT | 3-6 weeks
  Time Frame: Baseline and 3-6 weeks post-ADT initiation Description: PSMA-PET scans performed at 3 or 6 weeks after ADT will be compared to baseline scans to identify newly visible lesions. The outcome will be reported as the number and proportion of participants with new lesions. Descriptive statistics will be used to summarize findings.
Establish the optimal duration of ADT necessary to achieve castrate level of testosteroneTime to castration-level testosterone (≤50 ng/dL) following initiation of oral ADT (relugolix 120 mg daily) | 3-6 weeks
  Time Frame: 0 to 6 weeks after initiation of ADT Description: Serum testosterone will be measured at baseline, 3 weeks, and 6 weeks. The time point at which testosterone ≤50 ng/dL is first achieved will be recorded for each participant. Data will be summarized by frequency, proportion, and median time to castration levels.
Proportion of lesions visible on baseline PSMA-PET that remain detectable on post-ADT PSMA-PET | 3-6 weeks
  Time Frame: Baseline and 3-6 weeks after initiation of ADT Description: Lesions identified at baseline will be matched to post-ADT PSMA-PET scans. The number and proportion of lesions that remain visible after ADT will be recorded. This will help assess whether ADT obscures PSMA-positive disease on imaging.

SECONDARY OUTCOMES:
Correlation between PSMA-PET findings and surgical pathology | 3-6 weeks
  Time Frame: Surgery performed 6-10 weeks after enrollment Description: Lesions identified by PSMA-PET will be compared to histopathologic findings from prostatectomy and pelvic lymph node dissection specimens. Correlation statistics (e.g., sensitivity, specificity, positive predictive value) will be calculated.
Concordance between study PSMA-PET and conventional imaging or alternative PSMA-PET agents (if available) | 3-6 weeks
  Time Frame: 3-6 weeks after ADT, when comparator imaging is available Description: In participants who undergo additional imaging (e.g., bone scan, CT, or alternative PSMA-PET tracers), lesions will be compared to those seen on study PSMA-PET. Concordance will be reported as number and proportion of lesions detected by both modalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Clinics of North Texas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://urologyclinics.com/clinicaltrials